CLINICAL TRIAL: NCT05253937
Title: Impact of Intracoronary Versus Central and Peripheral Intravenous Epinephrine Administration During Cardiac Arrest in The Cardiac Catheterization Laboratory for Acute Myocardial Infarction Patients.
Brief Title: Impact of Intracoronary Versus Intravenous Epinephrine Administration During Cardiac Arrest .
Acronym: (iCPR)
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Baylor Scott and White Health (Other); Minneapolis Heart Institute (Other)
Responsible Party: Principal Investigator, Ali Aldujeli, Cardiovascular disease consultant, Lithuanian University of Health Sciences
Other Study IDs: LUHSKC-175
Record Dates: First submitted 2022-01-23; First posted 2022-02-24 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Cardiopulmonary Arrest; Epinephrine Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Heart Arrest | interventions — Epinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intracoronary Epinephrine administration during cardiac arrest
  Interventions: Drug: Epinephrin
- Peripheral intravenous Epinephrine administration during cardiac arrest
  Interventions: Drug: Epinephrin
- Central intravenous Epinephrine administration during cardiac arrest
  Interventions: Drug: Epinephrin

INTERVENTIONS:
Drug: Epinephrin — The study will enroll acute myocardial infarction patients who suffered from a cardiac arrest in the cardiac catheterization laboratory during percutaneous intervention procedure. Cardiac Resuscitation was performed according to the European Resuscitation Council (ERC) Guidelines. The preferred route of epinephrine administration was through the central venous access (by internal jugular or subclavian vein). Thus, if available, it was the preferred method of medication delivery. However, in cases without central venous access, the route of epinephrine administration (peripheral intravenous or arterial intracoronary) during cardiac arrest was left to the treating physicians.

SUMMARY:
In hospital cardiac arrest (IHCA) is a major challenge imposed on almost all health care systems worldwide. Despite significant progress in cardiopulmonary resuscitation in the past few years, outcomes remain relatively poor with an approximate 49 % survival rate.

Epinephrine administration remains a cornerstone in the treatment of cardiac arrest. However, the preferred route of administration remains a matter of debate within the medical community .

Various routes of administration, including intravenous, intramuscular, intraosseous and endotracheal routes have been studied.

Initially, American guidelines for the treatment of cardiac arrest recommended injection of 0.5 mg of epinephrine directly into the right ventricle through the parasternal approach, aiming to achieve higher peak intracardiac concentrations and a more central effect, however the intravenous route remained preferable due to its feasibility and safety .

To our knowledge, intra-coronary epinephrine administration for intraprocedural cardiac arrest has not been evaluated or compared with other routes of administration.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years old
* Diagnosed with non-ST elevation myocardial infarction (NSTEMI) or ST elevation myocardial infarction (STEMI)
* Received dual antiplatelet therapy (acetylsalicylic acid and ticagrelor), or triple therapy (oral anticoagulant, acetylsalicylic acid and clopidogrel)
* Event of cardiac arrest during percutaneous intervention

Exclusion Criteria:

* cardiac arrest documented prior to being transported to cardiac catheterization laboratory.
* Patients who suffered cardiac arrest for less than 60 seconds were excluded from the study.
* Received mechanical circulatory support such as intra-aortic balloon pump, temporary percutaneous ventricular assist devices, or extracorporeal membrane oxygenation (ECMO) during hospitalization.
* Presenting with any cardiac rhythm on admission other than sinus rhythm or atrial fibrillation/flutter
* Signs of infection or a history of hepatic, oncologic or allergy to contrast media and end stage renal failure
* Patients who underwent primary fibrinolysis.
* Furthermore, patients who received atropine, amiodarone, lidocaine, or any other antiarrhythmic prior to CPR
* who received targeted temperature management post CPR .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective, cohort, dual center pilot study, conducted in the Hospital of the Lithuanian University of Health Sciences Kaunas Clinics and the Republican Hospital of Panevezys from 2018 to 2022. Both cardiac centers covers six out of ten administrative regions in the republic of Lithuania.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
ROSC (return of spontaneous circulation) between different routes of epinephrine administration. | Up to 24 hours
  Return of sinus rhythm or atrial fibrillation/flutter for more than 5 minutes (through ECG monitoring)

SECONDARY OUTCOMES:
Survival to hospital discharge with favorable neurologic status (CPC score1-2) | Up to 30 days
  Cerebral Performance Category (CPC) - a five point scale that ranges from good cerebral performance (1) to brain death (5), is often used and is commonly dichotomized into "good" (CPC 1-2) versus "poor" (CPC 3-5) outcome .

OTHER OUTCOMES:
inhospital stent thrombosis | Up to 30 days
  Stent thrombosis confirmed by diagnostic angiography or sudden ST elevation on ECG in the specific segments confounding with stent location

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Aldujeli, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aldujeli A, Haq A, Tecson KM, Kurnickaite Z, Lickunas K, Bailey S, Tatarunas V, Braukyliene R, Baksyte G, Aldujeili M, Khalifeh H, Briedis K, Ordiene R, Unikas R, Hamadeh A, Brilakis ES. A prospective observational study on impact of epinephrine administration route on acute myocardial infarction patients with cardiac arrest in the catheterization laboratory (iCPR study). Crit Care. 2022 Dec 20;26(1):393. doi: 10.1186/s13054-022-04275-8. PMID 36539907